CLINICAL TRIAL: NCT01056952
Title: Physiologic Effects of High Flow Nasal Therapy in Patients With Acute Hypoxemic Respiratory Failure
Brief Title: Physiologic Effects of High Flow Nasal Therapy in Patients With Acute Hypoxemic Respiratory Failure (OPTIFLOW)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2009/15
Record Dates: First submitted 2010-01-18; First posted 2010-01-26 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optiflow then CPAP (Experimental): Standard low flow oxygen therapy then High flow oxygen nasal therapy (Optiflow)then Continuous positive airway pressure (CPAP)
  Interventions: Procedure: O2stand; Procedure: CPAP; Procedure: Optiflow
- CPAP then Optiflow (Experimental): Standard low flow oxygen therapy then Continuous positive airway pressure (CPAP)then High flow oxygen nasal therapy (Optiflow)
  Interventions: Procedure: O2stand; Procedure: CPAP; Procedure: Optiflow

INTERVENTIONS:
Procedure: O2stand — Standard low flow oxygen therapy (O2stand). The patients will receive oxygen delivered through a face mask. The FiO2 will be adjusted in order to obtain a SaO2 > 90%. The FiO2 will be determined by a portable oxygen analyzer (MiniOX I; Mine Safety Appliances Co, Pittsburgh, Pa)
Procedure: CPAP — o Continuous positive airway pressure (CPAP). CPAP will be set at 7.5 cmH2O. Airway humidification will be achieved by using a heated humidifier (MR640; Fisher & Paykel, Auckland, NZ). The FiO2 will be adjusted in order to obtain a SaO2 > 90%. A facial mask composed of a transparent mask and a soft inflatable will be used
Procedure: Optiflow — High flow oxygen nasal therapy (Optiflow). The flow will be set at 40l/min. The inspired fraction of oxygen (FiO2) will be adjusted in order to obtain a SaO2 > 90%

SUMMARY:
The aim of the study is to assess, in patients with acute hypoxemic respiratory failure, the short term physiologic effects of the high flow oxygen nasal therapy (Optiflow), in term of inspiratory muscle effort, gas exchange, comfort and dyspnea

DETAILED DESCRIPTION:
The administration of a known concentration of oxygen is an important part of routine care of the patient admitted in intensive care unit for acute hypoxemic respiratory failure. A new high flow oxygen delivery system (Fisher and Paykel Health care) has been developed (Optiflow). The system used a heated humidifier and heated breathing circuit via a nasal interface. High flow nasal therapy (Optiflow) is associated with the generation of significant positive airway pressure in healthy volunteers. Positive expiratory pressure may have a number of benefits in respiratory failure which include improved ventilation/perfusion matching with improved oxygenation, reduced airways resistance and reduced work of breathing. Moreover high flow nasal therapy may improve oxygen administration by decreasing oxygen dilution, decreasing death space and using high levels of humidification

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory insufficiency, defined as the PaO2/FIO2 ratio of 300 mm Hg or less after breathing oxygen
* The presence of lung infiltrates on a posteroanterior chest radiograph

Exclusion Criteria:

* Face or cranial trauma or surgery
* Patients younger than 18 years
* History of COPD
* Acute respiratory acidosis (defined as a pH <7.30 and a PaCO2 >50 mm Hg)
* Hemodynamic instability with arterial pressure < 90mmHg
* Respiratory instability with PaO2/FiO2<100mmHg
* ventricular arrhythmias
* Excess respiratory secretions.
* Upper gastrointestinal bleeding
* Recent gastric or oesophageal surgery
* Tracheostomy or other airways disorders
* Pneumothorax
* Contraindication of gastric probe insertion
* Impossibility to insert the oesophageal probe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle effort : oesophageal pressure (Poes) and the oesophageal pressure time product (PTPoes) | Every 30 minutes for 90 minutes

SECONDARY OUTCOMES:
Gas exchange :PaO2/FiO2 ratio | Every 30 minutes for 90 minutes
Comfort assessed using a five-item semi quantitative scale | Every 30 minutes for 90 minutes
Dyspnea assessed using a visual analogic scale | Every 30 minutes for 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric VARGAS, MD, Principal Investigator — University Hospital, Bordeaux, France
Locations (1):
- Pellegrin Hospital, Recovery Unit, Bordeaux, France

REFERENCES:
- [Derived] Vargas F, Saint-Leger M, Boyer A, Bui NH, Hilbert G. Physiologic Effects of High-Flow Nasal Cannula Oxygen in Critical Care Subjects. Respir Care. 2015 Oct;60(10):1369-76. doi: 10.4187/respcare.03814. Epub 2015 May 5. PMID 25944940